CLINICAL TRIAL: NCT00606619
Title: Phase III Clinical Trial for Effect Early Oral Feeding on Recovery After Resection of Gastric Cancer
Brief Title: Effects of Early Oral Feeding After Resection of Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Hae Myung Jeon, MD, Department of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCMC07OT135
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-02

CONDITIONS: Gastric Cancer
Keywords: Gastrectomy; Oral feeding; Nutrition; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Conventional feeding : They begin ingesting sips of water on third postoperative day and continued with a liquid diet for the next two days. Patients were given a soft diet on sixth postoperative day.
  Interventions: Other: Conventional feeding
- 2 (Experimental): Early oral feeding : The patients begin ingesting sips of water on the first postoperative day. If they are tolerable, they continued with a clear liquid diet the next day and a soft diet on the third post operative day.
  Interventions: Other: Early oral feeding

INTERVENTIONS:
Other: Conventional feeding — Procedure of Conventional feeding group: Patients are supplied water on day 3 after operation, liquid diet on day 4 and 5 and soft diet on 6 day.
  Arms: 1
Other: Early oral feeding — Procedure of Early oral feeding group: Patients are supplied water on day 1 after operation, liquid diet on day 2 and soft diet on day 3 day.
  Arms: 2

SUMMARY:
The aim of this study is to determine whether early oral feeding after curative resection for gastric cancer would be tolerable and give an effect on the recovery.

DETAILED DESCRIPTION:
Most patients who undergo gastric resection for gastric cancer have maintained going on a fast of over three days after operation. Surgeons have believed that early oral feeding might worsen patients' condition by prolonged postoperative ileus. Therefore, patients received nothing by oral route until resolution of the ileus. However, the current trend toward minimal operative injury and early discharge from hospital. In addition, development of operative technique and instrument make the operation time to be short and the patients to be fast recovery, and thus it is possible to feed early in less than two days after operation. The aim of this study is to determine whether early oral feeding after curative resection for gastric cancer would be tolerable and give an effect on the recovery.

We collect fifty-eight patients for this study and divide into two groups using randomization method. In the early feeding group, patients will receive the liquid diet two day after operation followed by soft diet postoperative three day. Meanwhile, the patients who categorized into control group will start the liquid diet postoperative four day followed by soft diet postoperative six day. We evaluate the morbidity or mortality rate and laboratory findings. Of course, it is supposed to be same in amount of fluid and calories between two groups.

ELIGIBILITY:
Inclusion Criteria:

Patients who underwent gastrectomy for adenocarcinoma of stomach with following criteria:

1. Performed curative resection
2. Have The American Society of Anaesthesiologists (ASA) score of less than 3

Exclusion Criteria:

1. Patients who have simultaneously other cancer.
2. Patients who underwent gastric resection at past time.
3. Patients who have cancer with bleeding or perforation or obstruction.
4. Patients who have any injury to the pancreas capsule on operation.
5. Patients who get pregnancy.
6. Patients who are treating diabetics with Insulin.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Days of hospital stay after operation | within 30 days after operation
  We measure the length of hospital stay after operation

SECONDARY OUTCOMES:
Day of recovery of bowel sound and flatus: Evidence of recovery of bowel sound by physician's examination and Evidence of first flatus by question to patient | within 30 days after operation
  We measure the days of flatus within 30 days after operation
Laboratory findings after operation: Albumin, complete blood count, total cholesterol, cholinesterase and C-reactive protein are measured | 1,3,5 and 7 day after operation
Symptom of Patients: Question to patients about symptoms | before operation and 1,3,5,7 day after operation
Cost effectiveness: Total cost duration of hospitalization | within 30 days after admission
  We measure total cost from admission to discharge after operation
Quality of life: EORTC QLQ30, STO22 | 1,2 and 3 month after operation
Immunologic Outcomes : IL-1, IL-2, IL-6, IL-8, TNF-a will by measured by ELISA | before operation and 1,3,5,7 day after operation
Postoperative morbidity rate in hospital days: Clinically definite morbidity confirmed by physicians according to offered protocol | within 30 days after operation
  We observe the occurrence of morbidity after operation

CONTACTS AND LOCATIONS:
Overall Officials: Hae Myung Jeon, MD, Principal Investigator — Department of Surgery, St Mary's Hospital, The Catholic University of Korea; Hoon Hur, MD, Study Director — Department of Surgery, St Mary's Hospital, The Catholic University of Korea
Locations (1):
- St Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

REFERENCES:
- [Background] Suehiro T, Matsumata T, Shikada Y, Sugimachi K. Accelerated rehabilitation with early postoperative oral feeding following gastrectomy. Hepatogastroenterology. 2004 Nov-Dec;51(60):1852-5. PMID 15532842
- [Background] Gabor S, Renner H, Matzi V, Ratzenhofer B, Lindenmann J, Sankin O, Pinter H, Maier A, Smolle J, Smolle-Juttner FM. Early enteral feeding compared with parenteral nutrition after oesophageal or oesophagogastric resection and reconstruction. Br J Nutr. 2005 Apr;93(4):509-13. doi: 10.1079/bjn20041383. PMID 15946413
- [Background] Reissman P, Teoh TA, Cohen SM, Weiss EG, Nogueras JJ, Wexner SD. Is early oral feeding safe after elective colorectal surgery? A prospective randomized trial. Ann Surg. 1995 Jul;222(1):73-7. doi: 10.1097/00000658-199507000-00012. PMID 7618972
- [Derived] Hur H, Si Y, Kang WK, Kim W, Jeon HM. Effects of early oral feeding on surgical outcomes and recovery after curative surgery for gastric cancer: pilot study results. World J Surg. 2009 Jul;33(7):1454-8. doi: 10.1007/s00268-009-0009-3. PMID 19399550